CLINICAL TRIAL: NCT03090750
Title: What is the Effect of Using Aromatherapy to Reduce Anxiety in Patients Undergoing Invasive Radiologic Procedures?
Brief Title: Effects of Aromatherapy on Anxiety in Invasive Radiologic Procedure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-14-09B
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2018-03

CONDITIONS: Anxiety; Anxiety Preoperative
MeSH Terms: conditions — Anxiety Disorders | interventions — lavender oil; bergamot oil; Water

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lavender (Experimental): Lavender oil
  Interventions: Drug: Lavender Oil
- Bergamot (Experimental): Bergamot oil
  Interventions: Drug: Bergamot Oil
- Water (Placebo Comparator): Water
  Interventions: Other: Water

INTERVENTIONS:
Drug: Lavender Oil — Lavender essential oil applied to cotton ball (3 drops) and placed in a medicine cup on bedside table
  Other Names: Lavender essential oil; Lavender; Lavender flower oil; Lavendula angustifolia
  Arms: Lavender
Drug: Bergamot Oil — Bergamot essential oil applied to cotton ball (3 drops) and placed in a medicine cup on bedside table
  Other Names: Bergamot essential oil; Bergamot; Citrus bergamia
  Arms: Bergamot
Other: Water — Tap water applied to cotton ball (3 drops) and placed in a medicine cup on bedside table
  Arms: Water

SUMMARY:
The purpose of this study is to see if using aromatherapy (Lavender or Bergamot) will lower anxiety in patients having invasive Radiology procedures. First, the level of anxiety is assessed prior to the procedure using a questionnaire. Then, patients are given the aromatherapy treatment during the pre-procedure period. Then, the same questions are asked to determine how anxious the patient is after the aromatherapy and before going into the procedure room. After the procedure, patients are asked to evaluate the process of the study.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Myelogram or IR invasive procedure at investigative site

Exclusion Criteria:

* Incapable of giving informed consent
* Requiring pre-medication for scheduled procedure
* Allergy to lavender or bergamot
* Asthma (type of breathing related condition)
* COPD (Chronic Obstructive Pulmonary Disorder - breathing disease)
* Respiratory issues requiring oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Anxiety level of patients | Immediately prior to invasive radiologic procedure
  Assessed with Amsterdam Preoperative Anxiety and Information Scale

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Becker, PhD, Principal Investigator — Wake Forest University Health Sciences